CLINICAL TRIAL: NCT04866511
Title: Video Narrative Exposure Therapy (NET) With Children and Young People Who Witnessed Domestic Violence: A Naturalistic Single Case Study Series
Brief Title: Video NET With CYP Who Witnessed Domestic Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottinghamshire Healthcare NHS Trust (Other Government); Lincolnshire Partnership NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21003; 291108 (Other: IRAS)
Record Dates: First submitted 2021-04-22; First posted 2021-04-29 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Post-Traumatic Stress Disorder in Children; Post-Traumatic Stress Disorder in Adolescence; Post-Traumatic Stress Disorder Complex; Domestic Violence; Trauma, Psychological; Narrative Exposure Therapy
Keywords: post-traumatic stress; narrative exposure therapy; children and young people; domestic violence; case study series
MeSH Terms: conditions — Psychological Trauma | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: The study will adopt a Single Case Design (SCD) methodology, and specifically a naturalistic, sequential measurement, mixed-method AB design.
  SCDs are an idiographic method that allows for the analysis and interpretation of change at the level of the individual, rather the group. As such, SCDs typically aim to measure the change occurring in the individual's behaviour or symptoms by comparing the baseline, the intervention and the follow-up phases in terms of trends and variability (Parsonson & Baer, 1986). Furthermore, SCDs lend themselves to an in-depth exploration of process and outcome of therapy in applied settings, and, particularly when experimental, allows for drawing causal inferences about effectiveness. This is in line with the objectives of this study, which aims to answer questions about both outcomes and processes of change within NET.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NET intervention (Experimental): This study will follow a single case design and will involve delivering and evaluating the child-friendly protocol of NET. Therefore, there will only be one arm (NET intervention) and no comparators.
  Interventions: Other: Narrative Exposure Therapy

INTERVENTIONS:
Other: Narrative Exposure Therapy — NET is a trauma-focused psychological treatment for people who experienced multiple traumas (Schaeur et al., 2011).
  An adaptation named KIDNET was developed for use with children and young people (Neuner et al., 2008; Schauer et al., 2011, 2017).
  Participants will be offered 6-10 weekly sessions of NET lasting approximately 90 minutes each. The sessions will be delivered by a Trainee Clinical Psychologist via videoconferencing, in line with the UK's Government guidelines around reducing face-to-face contacts during the Covid-19 pandemic.
  Other Names: NET; KIDNET (protocol for children and adolescents)

SUMMARY:
Research suggests that children and young people (CYP) who witness domestic violence are susceptible to develop Post-traumatic stress (PTS). As their traumatic experiences are often repeated and prolonged, these CYP are likely to present with 'complex trauma' presentations, which also include other difficulties such as depressive symptoms and problems in functioning.

This study aims to investigate whether Narrative Exposure Therapy (NET) delivered via videoconferencing can be effective, feasible, and acceptable for CYP who witnessed domestic violence. NET is a brief, evidence-based intervention for complex trauma which has been adapted for CYP. The study will use a 'single case study series' design and look at whether NET can impact on PTS, psychological distress, and functioning. It will also look at the processes of change within NET and participants' experience of the therapy. Young people aged 12-17 who are experiencing PTS after exposure to domestic violence will be recruited from the waiting lists of Child and Adolescent Mental Health Services in Lincolnshire Partnership NHS Foundation Trust and Nottinghamshire Healthcare NHS Foundation Trust.

Up to six participants will receive six to ten weekly video sessions and the changes in the outcomes will be explored before, during and after NET. Finally, participants will be interviewed about their experiences.

The study is part of a Doctorate in Clinical Psychology programme and funded by Health Education England. Potential benefits include investigating NET with a new group, contributing to the research on complex trauma interventions for CYP, and providing insights on the effectiveness and acceptability of therapies via video.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the potential effectiveness, feasibility, acceptability and putative mechanisms of change of video NET with children and young people who witnessed domestic violence.

The primary objective of the study is to evaluate whether video NET can reduce PTS in this group.

The secondary objectives of the study are:

* To determine whether video NET can also impact on general psychological distress and functioning;
* To examine the putative mechanisms of change within NET, i.e. habituation and integration of trauma memories;
* To explore the feasibility and acceptability of video NET.

ELIGIBILITY:
Inclusion Criteria - Participants must:

* Be aged 12- 17;
* Have witnessed domestic violence in the past;
* Be experiencing clinical levels of post-traumatic stress, as assessed by a member of the CAMHS team;
* Be on the waiting list to receive trauma-focused treatment;
* If 16 or over, be able to consent to take part, as assessed by a member of the CAMHS team;
* If under 16, have at least one person with parental authority who can consent for them. These young people will also be asked to provide their assent;
* Be able to communicate verbally and speak English;
* Have access to a device with a webcam and Internet broadband to enable participation in video sessions;
* Have access to a mobile device, e.g. a smartphone or a tablet. Can be the same as the device above.

Exclusion Criteria - Participants will be excluded from the study if:

* They have a known diagnosis of Intellectual Disability;
* They have a current high level of risk including of self-harm, suicide or current exposure to domestic violence, as assessed by a member of the CAMHS team;
* They are substance dependent.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Change in PTS symptoms between the baseline, NET intervention, and 1-month follow-up phases - as assessed by the Children's Revised Impact of Event Scale (CRIES-13; Perrin et al., 2005) | Throughout the study, for approximately 18 weeks
  The CRIES is a brief self-report questionnaire assessing PTS in children and young people aged 8-18. The original version of the scale (CRIES-8) includes 8 items evaluating intrusion and avoidance symptoms; a longer version (CRIES-13) comprising 5 additional items was developed to include the assessment of hyperarousal symptoms. The young person completing the scale is asked to rate each item depending on how frequently they experienced the symptom in the past week on a four-point scale . Although the CRIES is not a diagnostic instrument, higher scores suggest higher levels of PTS and likely clinical caseness. The scale has demonstrated good face and construct validity and has been used to screen and capture symptom change in children exposed to a variety of traumatic events (Perrin et al., 2005; Smith et al., 2003).

SECONDARY OUTCOMES:
Change in pyschological distress and functioning between the baseline, NET intervention, and 1-month follow-up phases - as assessed by the Young Person's Clinical Outcomes in Routine Evaluation (YP-CORE; Twigg et al., 2009) | Throughout the study, for approximately 18 weeks
  The YP-CORE has been adapted from the CORE-10 for use with children and young people between 11 and 16 years. The scale is a session-by-session monitoring tool comprising items assessing anxiety symptoms, depression symptoms, physical problems, functioning and risk to self. The YP-CORE includes six high severity items and four low severity items. When completing the YP-CORE, the young person rates the 10 items based on how often they experienced each problem over the past week (0 = "Not at all", 1 = "Only occasionally", 2 = "Sometimes", 3 = "Often", 4 = "Most or all of the time"). Previous studies have demonstrated the scale's reliability, validity and sensitivity to change (Twigg et al., 2009; Twigg et al., 2016).

OTHER OUTCOMES:
Process measure of habituation: Heart Rate (HR) wristband monitor | For approximately 10 weeks
  HR monitors have been recommended for use as a proxy measure of physiological arousal (Schäfer et al., 2018). In the proposed study, changes in HR will be used to measure: a) within-session habituation (WSH) before and after exposure to traumatic narratives; b) and between-session habituation (BSH) as the narration progresses. Commercially available monitors include chest straps and wristbands; the latter type was deemed less invasive for participants and thus chosen for this study. Huawei Band 4 Pro is an example of a wearable activity tracker that includes a continuous heart rate monitor function. The product can be connected with the manufacturer's app (Huawei Health) installed on an Android or IOS mobile device.
Process measure of integration of trauma memories: Trauma Memory Quality Questionnaire (TMQQ; Meiser-Stedman et al. 2007) | Approximately 10 weeks
  The TMQQ is an 11-item self-report questionnaire designed to assess the problematic characteristics of traumatic memories resulting from a lack of autobiographical integration (e.g. fragmentation, sensory/visual rather than verbal quality etc.) in children and young people. The young person rates the item on a 4-point scale (1 = "Don't agree at all", 2 = "Don't agree a bit", 3 = "Agree a bit", 4 = "Completely agree") how well the statements reflect their trauma memories. Higher scores are indicative of more problematic and less integrated memories. The scale has been previously employed to measure the impact of NET on the quality of traumatic memories (Peltonen & Kangaslampi, 2019; Isoaho et al., 2015).
Change interviews | At 1-month follow-up
  The feasibility and acceptability of video NET will be investigated by conducting Change Interviews with the young people approximately one month after completing the treatment. In this instance, the young people will also be asked to provide feedback on their experience of receiving treatment via videoconferencing, including in terms of barriers and fascinators to engagement. The interviews will be conducted by an external researcher, i.e. another Trainee Clinical Psychologist, following an adaptation of Elliott, Slatick, & Urman's (2001) protocol. The interviews will be audio- or video-recorded and then sent to the student/investigator for transcription and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schröder, PhD, Study Director — University of Nottingham; Sarah Wilde, DClinPsy, Study Director — University of Lincoln; Fiammetta Rocca, Trainee Clinical Psychologist, MSc, Principal Investigator — University of Nottingham; Nima Moghaddam, PhD, DClinPsy, Study Director — University of Lincoln
Locations (2):
- United Kingdom (2):
  - Lincolnshire Partnership Foundation NHS Trust - Child and Adolescent Mental Health Services, Lincoln, Lincolnshire
  - Nottinghmashire Healthcare NHS Foundation Trust - Community Child and Adolescent Mental Health Services, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neuner F, Catani C, Ruf M, Schauer E, Schauer M, Elbert T. Narrative exposure therapy for the treatment of traumatized children and adolescents (KidNET): from neurocognitive theory to field intervention. Child Adolesc Psychiatr Clin N Am. 2008 Jul;17(3):641-64, x. doi: 10.1016/j.chc.2008.03.001. PMID 18558317
- [Background] Schauer, M., Neuner, F., & Elbert, T. (2011). Narrative exposure therapy: A short-term treatment for traumatic stress disorders (2nd rev. and expanded ed.). Hogrefe Publishing.
- [Background] Schauer, M., Neuner, F., & Elbert, T. (2017). Narrative Exposure Therapy for Children and Adolescents (KIDNET). In M. A. Landolt, M. Cloitre, & U. Schnyder (Eds.), Evidence-Based Treatments for Trauma Related Disorders in Children and Adolescents (pp. 227-250). Springer.
- [Background] Parsonson, B. S., & Baer, D. M. (1986). The graphic analysis of data. In J. S. Bailey & M. R. Burch (Eds.), Research methods in applied behavior analysis (pp. 157-186). Springer.
- [Background] Perrin, S., Meiser-Stedman, R., & Smith, P. (2005). The Children's Revised Impact of Event Scale (CRIES): Validity as a screening instrument for PTSD. Behavioural and Cognitive Psychotherapy, 33(4), 487-498.
- [Background] Twigg, E., Barkham, M., Bewick, B. M., Mulhern, B., Connell, J., & Cooper, M. (2009). The Young Person's CORE: Development of a brief outcome measure for young people. Counselling and Psychotherapy Research, 9(3), 160-168.
- [Background] Twigg E, Cooper M, Evans C, Freire E, Mellor-Clark J, McInnes B, Barkham M. Acceptability, reliability, referential distributions and sensitivity to change in the Young Person's Clinical Outcomes in Routine Evaluation (YP-CORE) outcome measure: replication and refinement. Child Adolesc Ment Health. 2016 May;21(2):115-123. doi: 10.1111/camh.12128. Epub 2015 Nov 3. PMID 32680371
- [Background] Schafer SK, Ihmig FR, Lara H KA, Neurohr F, Kiefer S, Staginnus M, Lass-Hennemann J, Michael T. Effects of heart rate variability biofeedback during exposure to fear-provoking stimuli within spider-fearful individuals: study protocol for a randomized controlled trial. Trials. 2018 Mar 16;19(1):184. doi: 10.1186/s13063-018-2554-2. PMID 29548298
- [Background] Meiser-Stedman R, Smith P, Yule W, Dalgleish T. The Trauma Memory Quality Questionnaire: preliminary development and validation of a measure of trauma memory characteristics for children and adolescents. Memory. 2007 Apr;15(3):271-9. doi: 10.1080/09658210701256498. PMID 17454664
- [Background] Peltonen K, Kangaslampi S. Treating children and adolescents with multiple traumas: a randomized clinical trial of narrative exposure therapy. Eur J Psychotraumatol. 2019 Jan 17;10(1):1558708. doi: 10.1080/20008198.2018.1558708. eCollection 2019. PMID 30693077
- [Background] Isoaho, P., Kangaslampi, S., & Peltonen, K. (2015). Narratiivisen altistusterapian (NET) vaikutus kognitiivisiin prosesseihin ja mielenterveyteen: Tapaustutkimus = The effect of Narrative Exposure Therapy (NET) on cognitive processes and mental health: A case study. Psykologia, 50(5), 355-372. https://proxy.library.lincoln.ac.uk/login?url=https://search.ebscohost.com/login.aspx?direct=true&db=psyh&AN=2015-52491-003&site=ehost-live
- [Background] Elliott, R., Slatick, E., & Urman, M. (2001). Qualitative Change Process Research on Psychotherapy: Alternative Strategies. Psychologische Beitrage, 43(3), 69-111.
- [Derived] Rocca F, Schroder T, Golijani-Moghaddam N, Wilde S. Video Narrative Exposure Therapy (NET) with Children and Young People who Witnessed Domestic Violence: A Naturalistic Single Case Study Series. J Child Adolesc Trauma. 2025 Jan 10;18(2):447-465. doi: 10.1007/s40653-024-00681-y. eCollection 2025 Jun. PMID 40469793